CLINICAL TRIAL: NCT03992417
Title: A Prospective Observational Study of Patients Receiving Dupixent® for Atopic Dermatitis
Brief Title: Observational Study of Patients Receiving Dupixent® for Atopic Dermatitis (AD)
Acronym: GLOBOSTAD
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS15990
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with AD: Adult and adolescent participants with AD initiating treatment with Dupixent® for AD according to the country-specific prescribing information, as part of their usual care as determined by their physician
  Interventions: Drug: Dupilumab SAR231893 (REGN668)

INTERVENTIONS:
Drug: Dupilumab SAR231893 (REGN668) — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous injection
  Other Names: Dupixent®

SUMMARY:
Primary Objective:

To characterize the patients who receive Dupixent® (dupilumab) for AD in a real-world setting, with respect to their medical history, socio-demographic and disease characteristics, and prior and concomitant treatments of AD

Secondary Objectives:

* To characterize real-world use patterns of Dupixent® for AD (eg, used regimens, reason for initiation of new treatments, concomitant therapies, treatment durations and reasons for discontinuation and/or switching)
* To assess the long-term effectiveness of Dupixent® in AD patients in a real-world setting
* To assess comorbid atopic conditions and effects of treatment in comorbid atopic conditions in patients who receive Dupixent® for AD
* To collect safety data on study participants

DETAILED DESCRIPTION:
Participants enrolled in the study will be followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 12 years or older at the baseline visit. Note: Adolescent participants (at least 12 years old, but less than 18 years) are eligible only after Dupixent® receives the respective country's regulatory approval for use in this age group;
* Initiating treatment with Dupixent® for AD according to the country-specific prescribing information. Note: Participants may be eligible if they have already initiated treatment with Dupixent® for AD within 6 months before their enrollment in the registry, provided that all core baseline data required (Eczema Area and Severity Index [EASI], Scoring of Atopic Dermatitis [SCORAD], body surface area [of AD involvement] [BSA], Patient-Oriented Eczema Measure [POEM], and Dermatology Life Quality Index [DLQI]) by the registry protocol were captured at the time of initiating Dupixent® treatment and are available for entry in the registry database
* Able to understand and complete study-related questionnaires
* Provide signed informed consent or parental/legally acceptable representative consent and/or patient assent where applicable

Exclusion Criteria:

* Participants who have a contraindication to the drug according to the country-specific prescribing information label
* Any condition that, in the opinion of the investigator, may interfere with patient's ability to participate in the study, such as short life expectancy, substance abuse, severe cognitive impairment, or other co-morbidities that can predictably prevent the participant patient from adequately completing the schedule of visits and assessments
* Patients currently participating in any interventional clinical trial which modifies patient care
* Prior use of Dupixent® within 6 months of the screening visit, or within 6 months of the baseline visit if screening and baseline occur on the same day

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population is adult and adolescent patients (male or female, ≥12 years old), who are initiating treatment with Dupixent® for AD according to the country-specific prescribing information.
Sampling Method: Non-Probability Sample
Enrollment: 955 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Baseline Characteristics: Medical history | Baseline to Month 60
Baseline Characteristics: Socio-demographics | Baseline to Month 60
Baseline Characteristics: Disease characteristics | Baseline to Month 60

SECONDARY OUTCOMES:
Physician Assessment: Body Surface Area Affected (BSA) by Atopic Dermatitis | Baseline to Month 60
  Percentage of BSA affected by AD assessed for each major section of the body
Physician Assessment: Eczema Area and Severity Index (EASI) | Baseline to Month 60
  Measure used in clinical practice and clinical trials to assess the severity and extent of AD
Physician Assessment: Scoring of Atopic Dermatitis (SCORAD) | Baseline to Month 60
  Measure used in clinical practice and clinical trials to standardize the evaluation of the severity and extent of AD
Participant Assessment: Patient Oriented Eczema Measure (POEM) | Baseline to Month 60
  Questionnaire used in clinical practice and clinical trials to assess disease symptoms in children and adults
Participant Assessment: Pruritus Numerical Rating Scale (NRS) | Baseline to Month 60
  Individual NRS used to rate the intensity of pruritus using a 0 to 10 numeric rating scale
Participant Assessment: Skin Pain or Soreness NRS | Baseline to Month 60
  Individual NRS used to rate skin pain and soreness using a 0 to 10 NRS
Participant Assessment: Skin Feeling Hot NRS | Baseline to Month 60
  Individual NRS used to rate the sensation of skin feeling hot (burning sensation) using a 0 to 10 NRS
Participant Assessment: Skin Sensitivity NRS | Baseline to Month 60
  Individual NRS used to rate skin sensitivity using a 0 to 10 NRS
Participant Assessment: Sleep Disturbance NRS | Baseline to Month 60
  Individual NRS used to report the severity of their sleep disturbance using a 0 to 10 NRS
Participant Assessment: Dermatology Life Quality Index (DLQI) for adults and Children Dermatology Life Quality Index (CDLQI) for adolescents | Baseline to Month 60
  Questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL)
Participant Assessment: Juniper Asthma Control Questionnaire (ACQ-5) | Baseline to Month 60
  Questionnaire to evaluate asthma control in participants with comorbid asthma
Participant Assessment: Allergic Rhinitis-Visual Analog Scale (AR-VAS) | Baseline to Month 60
  Instrument for the documentation of symptoms and therapy monitoring in allergic rhinitis
Participant Assessment: Work Productivity and Activity Impairment Questionnaire for AD (WPAI-AD) for adults and Work Productivity and Activity Impairment Questionnaire+Classroom Impairment Questions for AD (WPAI-CIQ-AD) for adolescents | Baseline to Month 60
  Questionnaire to assess the impact of AD on productivity
Participant Assessment: Health Care Resource Utilization Questionnaire | Baseline to Month 60
  Questionnaire regarding hospitalization, or emergency room/urgent care center visits due to AD
Participant Assessment: 9-Item Treatment Satisfaction Questionnaire for Medication (TSQM-9) | Baseline to Month 60
  Instrument to measure treatment satisfaction
Adverse events (AEs) | Baseline to Month 60
  Number of participants with at least 1 AE
Participant Assessment: Atopic Dermatitis Control Tool (ADCT) to be collected optionally | Baseline to Month 60
  Questionnaire related with Atopic dermatitis control

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (114):
- Argentina (3):
  - Investigational Site Number : 0320013, Pilar, Buenos Aires
  - Investigational Site Number : 0320012, Rosario, Santa Fe Province
  - Investigational Site Number : 0320011, Ciudad Autonoma Bs As
- Australia (5):
  - Investigational Site Number : 0360002, Kogarah, New South Wales
  - Investigational Site Number : 0360005, Kogarah, New South Wales
  - Investigational Site Number : 0360003, Woolloongabba, Queensland
  - Investigational Site Number : 0360004, Bedford Park, South Australia
  - Investigational Site Number : 0360001, Carlton, Victoria
- Austria (4):
  - Investigational Site Number : 0400005, Graz
  - Investigational Site Number : 0400004, Linz
  - Investigational Site Number : 0400002, Maria Enzersdorf
  - Investigational Site Number : 0400001, Vienna
- Belgium (8):
  - Investigational Site Number : 0560002, Brussels
  - Investigational Site Number : 0560007, Edegem
  - Investigational Site Number : 0560010, Ghent
  - Investigational Site Number : 0560003, Jette
  - Investigational Site Number : 0560001, Leige
  - Investigational Site Number : 0560008, Leuven
  - Investigational Site Number : 0560004, Namur
  - Investigational Site Number : 0560006, Roeselare
- Colombia (3):
  - Investigational Site Number : 1700008, Bogotá
  - Investigational Site Number : 1700012, Bogotá
  - Investigational Site Number : 1700011, Medellín
- Czechia (7):
  - Investigational Site Number : 2030008, Hradec Králové
  - Investigational Site Number : 2030006, Olomouc
  - Investigational Site Number : 2030003, Ostrava - Poruba
  - Investigational Site Number : 2030004, Pilsen
  - Investigational Site Number : 2030005, Prague
  - Investigational Site Number : 2030002, Prague
  - Investigational Site Number : 2030001, Ústí nad Labem
- Investigational Site Number : 2460002, Kokkola, Finland
- France (9):
  - Investigational Site Number : 2500011, Antony
  - Investigational Site Number : 2500004, Auxerre
  - Investigational Site Number : 2500003, Bordeaux
  - Investigational Site Number : 2500009, Montpellier
  - Investigational Site Number : 2500006, Pierre-Bénite
  - Investigational Site Number : 2500010, Rouen
  - Investigational Site Number : 2500005, Saint-MandÃ© Cedex
  - Investigational Site Number : 2500002, Toulouse
  - Investigational Site Number : 2500001, Valence
- Greece (3):
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000003, Thessaloniki
  - Investigational Site Number : 3000001, Thessaloniki
- Israel (6):
  - Investigational Site Number : 3760006, Afula
  - Investigational Site Number : 3760005, Haifa
  - Investigational Site Number : 3760001, Haifa
  - Investigational Site Number : 3760002, Jerusalem
  - Investigational Site Number : 3760004, Ramat Gan
  - Investigational Site Number : 3760003, Rehovot
- Italy (15):
  - Investigational Site Number : 3800009, Torrette Di Ancona, Ancona
  - Investigational Site Number : 3800017, Terracina, Latina
  - Investigational Site Number : 3800003, Rome, Roma
  - Investigational Site Number : 3800011, Rome, Roma
  - Investigational Site Number : 3800012, Bari
  - Investigational Site Number : 3800007, Brescia
  - Investigational Site Number : 3800013, Cagliari
  - Investigational Site Number : 3800008, Genova
  - Investigational Site Number : 3800015, L’Aquila
  - Investigational Site Number : 3800004, Milan
  - Investigational Site Number : 3800001, Napoli
  - Investigational Site Number : 3800018, Palermo
  - Investigational Site Number : 3800010, Pisa
  - Investigational Site Number : 3800005, Roma
  - Investigational Site Number : 3800016, Torino
- Japan (16):
  - Investigational Site Number : 3920004, Nagakute-shi, Aichi-ken
  - Investigational Site Number : 3920015, Obihiro-shi, Hokkaido
  - Investigational Site Number : 3920006, Sapporo, Hokkaido
  - Investigational Site Number : 3920011, Hirakata-shi, Osaka
  - Investigational Site Number : 3920008, Koshigaya-shi, Saitama
  - Investigational Site Number : 3920005, Shimotsuga-gun, Tochigi
  - Investigational Site Number : 3920003, Itabashi-ku, Tokyo
  - Investigational Site Number : 3920022, Amagasaki-shi
  - Investigational Site Number : 3920002, Habikino-shi
  - Investigational Site Number : 3920014, Hamamatsu
  - Investigational Site Number : 3920025, Kyoto
  - Investigational Site Number : 3920013, Marugame-shi
  - Investigational Site Number : 3920012, Minokamo-shi
  - Investigational Site Number : 3920001, Nagoya
  - Investigational Site Number : 3920010, Setagaya-ku
  - Investigational Site Number : 3920020, Yokohama
- Investigational Site Number : 4140001, Sulaibikat, Kuwait
- Investigational Site Number : 4840001, Guadalajara, Jalisco, Mexico
- Investigational Site Number : 5280002, Bergen op Zoom, Netherlands
- Norway (2):
  - Investigational Site Number : 5780002, Bergen
  - Investigational Site Number : 5780001, BodÃ¸
- Portugal (4):
  - Investigational Site Number : 6200003, Coimbra
  - Investigational Site Number : 6200002, Lisbon
  - Investigational Site Number : 6200004, Porto
  - Investigational Site Number : 6200001, Vila Nova de Gaia
- Russia (3):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430002, Moscow
  - Investigational Site Number : 6430004, Saint Petersburg
- Saudi Arabia (2):
  - Investigational Site Number : 6820013, Dammam
  - Investigational Site Number : 6820001, Jeddah
- Spain (15):
  - Investigational Site Number : 7240019, Bilbao, Bizkaia
  - Investigational Site Number : 7240004, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number : 7240012, Majadahonda, Madrid
  - Investigational Site Number : 7240002, Oviedo, Principality of Asturias
  - Investigational Site Number : 7240011, Santullano de Mieres, Principality of Asturias
  - Investigational Site Number : 7240017, Barakaldo
  - Investigational Site Number : 7240009, Barcelona
  - Investigational Site Number : 7240014, Barcelona
  - Investigational Site Number : 7240021, Granada
  - Investigational Site Number : 7240016, Madrid
  - Investigational Site Number : 7240007, Madrid
  - Investigational Site Number : 7240006, Madrid
  - Investigational Site Number : 7240010, Madrid
  - Investigational Site Number : 7240001, Madrid
  - Investigational Site Number : 7240008, Santiago de Compostela
- Taiwan (4):
  - Investigational Site Number : 1580012, Kaohsiung City
  - Investigational Site Number : 1580011, Taichung
  - Investigational Site Number : 1580014, Taipei
  - Investigational Site Number : 1580015, Taoyuan
- Investigational Site Number : 7840002, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Calzavara-Pinton P, Chu CY, Lapeere H, Rossi M, Ferrucci SM, Chung WH, Fougerousse AC, Fomina DS, Holzer G, Celakovska J, Al-Ahmad M, Tzellos T, Wu J, Ardeleanu M, Bosman K. One-Year Insights into the GLOBOSTAD Multinational Prospective Observational Study of Patients Receiving Dupilumab for Atopic Dermatitis. Adv Ther. 2025 Feb;42(2):720-733. doi: 10.1007/s12325-024-03049-8. Epub 2024 Dec 2. PMID 39621227
- [Derived] Calzavara-Pinton P, Celakovska J, Lapeere H, Holzer G, Al-Ahmad M, Chu CY, Ferrucci SM, Kataoka Y, Rossi M, Fomina DS, Chung WH, Tzellos T, Fougerousse AC, Wu J, Ardeleanu M, Ozturk ZE. Baseline Demographics, Comorbidities, Treatment Patterns and Burden of Atopic Dermatitis in Adults and Adolescents from the GLOBOSTAD Long-Term Observational Study. Adv Ther. 2023 Dec;40(12):5366-5382. doi: 10.1007/s12325-023-02644-5. Epub 2023 Oct 6. PMID 37801232